CLINICAL TRIAL: NCT05019911
Title: Prediction of Exacerbations and Management of COPD Patients With Sleep Apnea Hypopnea Based on Millimeter Wave Radar Monitoring
Brief Title: Prediction of Exacerbations and Management of COPD Patients With SAH Based on Millimeter Wave Radar Monitoring
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Sponsor
Other Study IDs: M2021074
Record Dates: First submitted 2021-06-29; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-06

CONDITIONS: COPD; Sleep Apnea Hypopnea Syndrome; Acute Exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients with COPD alone: In the cross-sectional part, the group of patients with COPD alone will be monitored by traditional sleep monitoring equipment (polysomnography) and millimeter wave radar equipment. In the cohort part, this group of patients will be continuously monitored by millimeter wave radar equipment for vital signs combined with pulse oxygen saturation, end expiratory CO2 and other indicators continuously monitored.
  Interventions: Device: Polysomnography; Device: Millimeter wave radar equipment
- Patients with COPD combined with sleep apnea hypopnea syndrome: In the cross-sectional part, the group of patients with COPD combined with sleep apnea hypopnea syndrome will be monitored by traditional sleep monitoring equipment (polysomnography) and millimeter wave radar equipment. In the cohort part, this group of patients will be continuously monitored by millimeter wave radar equipment for vital signs combined with pulse oxygen saturation, end expiratory CO2 and other indicators continuously monitored.
  Interventions: Device: Polysomnography; Device: Millimeter wave radar equipment

INTERVENTIONS:
Device: Polysomnography — In the cross-sectional part, the group of patients with COPD alone and the group of patients with COPD combined with sleep apnea hypopnea syndrome will be monitored by traditional sleep monitoring equipment (polysomnography) for vital signs in order to diagnose COPD combined with sleep apnea hypopnea syndrome.
Device: Millimeter wave radar equipment — In the cross-sectional part, the group of patients with COPD alone and the group of patients with COPD combined with sleep apnea hypopnea syndrome will be monitored by millimeter wave radar equipment for vital signs in order to diagnose COPD combined with sleep apnea hypopnea syndrome. In the cohort part, both groups of patients will be continuously monitored by millimeter wave radar equipment for vital signs for months in order to establish a model to predict acute exacerbations of COPD combined with sleep apnea hypopnea syndrome.

SUMMARY:
Millimeter wave radar will be used to conduct non-contact monitoring continuously for patients' vital signs (eg. respiratory rate, heart rate, and chest/abdominal movement). The monitoring information will be transmitted to the central system through network and displayed in real time. Comparison with polysomnography will be done to examine the consistency between the two devices in diagnosing sleep breathing disorders. The predictive model of acute exacerbations of COPD will be established with the baseline indicators considered.

DETAILED DESCRIPTION:
Significance: This study will conduct non-contact monitoring among COPD patients with sleep apnea hypopnea for respiratory rate, heart rate, respiratory rhythm and thoracic amplitude. This monitoring could not only offer patients a more comfortable medical environment, but also maintain high quality of monitoring, which would help build the platform for prediction and management of COPD combined with sleep breathing disorders with great clinical significance.

Background: The misdiagnosis, underdiagnosis and disease burden of sleep breathing disorders in patients with COPD are high, which is one of the neglected problems in the management of COPD in China at present. The prevalence of obstructive sleep apnea (OSA) among COPD patients is 37.9-52.8%. Patients with overlapping COPD and OSA had more frequent hypoxemia during sleep and a longer total sleep duration for hypoxemia and hypercapnia than patients with OSA or COPD alone. The millimeter-wave radar equipment used in this study is from Qinglei Intelligent Health Care Life Support System. The system is based on millimeter wave radar intellisense and artificial intelligence technology, geared to the needs of health institutions, community endowment, family endowment, medical institutions, etc., to provide sleep monitoring, monitoring vital signs data, user behavior analysis, life vigor analysis, user exception alarm, falling alarm, diagnosis and screening of chronic respiratory disease, help with primary screening and early diagnosis of the disease and the patient-centered personalized precision diagnosis and treatment, enable early detection and treatment of health risks through scientific and technological means, and make more effective use of medical resources. The Peking University Third Hospital has actively promoted the construction of Internet-based medical services, and has passed the on-site evaluation of Internet hospital qualification, and realized Internet-based diagnosis and treatment. The Department of Respiratory and Critical Care Medicine has been engaged in clinical and applied basic research on COPD and its complications for a long time, which has a in-depth research foundation.

Objective: To verify the consistency between millimeter wave radar equipment and traditional sleep monitoring equipment in the collection of respiratory rate, heart rate and respiratory movement of patients with COPD alone or COPD combined with sleep apnea hypopnea syndrome. Combined with pulse oxygen saturation, end expiratory CO2 monitoring and other indicators, the data model established is conducive to early detection of aggravation of COPD combined with sleep apnea hypopnea syndrome based on clinical indicators, which has important clinical value in practice.

Content: Millimeter wave radar will be used to conduct non-contact monitoring continuously for patients' vital signs (eg. respiratory rate, heart rate, and chest/abdominal movement). The monitoring information will be transmitted to the central system through network and displayed in real time. Comparison with polysomnography will be done to examine the consistency between the two devices in diagnosing sleep breathing disorders. The predictive model of acute exacerbations of COPD will be established with the baseline indicators considered.

Methods: The patients with COPD alone and patients with COPD combined with sleep apnea hypopnea were monitored by traditional sleep monitoring equipment and millimeter wave radar equipment. The patients were continuously monitored by millimeter wave radar equipment and followed up for acute exacerbation of COPD.

Period: October 2021-September 2022 Expected results: The consistency between non-contact millimeter-wave radar equipment and routine clinical monitoring in the diagnosis of COPD combined with sleep apnea hypopnea syndrome. Based on the non-contact millimeter-wave radar equipment, a predictive model of acute exacerbation of COPD combined with sleep apnea hypopnea syndrome was established to provide evidence for the clinical application of radar equipment in the future.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD in line with Group on Chronic Obstructive Pulmonary disease, Chinese Thoracic Society. Guidelines for the diagnosis and treatment of chronic obstructive pulmonary disease (2013 revised).
* Or with Clinical diagnosis of sleep apnea hypopnea in line with Group on sleep breathing disorders, Chinese Thoracic Society. Guidelines for the diagnosis and treatment of obstructive sleep apnea hypopnea syndrome (2011 revised).
* Aged 40 years or older.
* Must provide informed consent.

Exclusion Criteria:

* Cognitive disorders.
* Unable to join in the study and so on.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD alone and patients with COPD combined with sleep apnea hypopnea syndrome aged 40 years or older
Sampling Method: Non-Probability Sample
Enrollment: 922 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index in times per hour | At baseline and millimeter wave radar monitoring continues during one month's or one year's follow-up
  AHI will be calculated by dividing times of apnea and hypopnea by hours of evaluation period during sleep.
  AHI will be monitored by millimeter wave radar devices and polysomnography.
Oxygen saturation in percent | At baseline and millimeter wave radar monitoring and pulse oximeter continues during one month's or one year's follow-up
  Oxygen saturation will be monitored by millimeter wave radar devices, polysomnography or pulse oximeter.
Respiratory rate in breaths per minute | At baseline and millimeter wave radar monitoring continues during one month's or one year's follow-up
  Respiratory rate will be monitored by millimeter wave radar devices and polysomnography.
Heart rate in beats per minute | At baseline and millimeter wave radar monitoring continues during one month's or one year's follow-up
  Heart rate will be monitored by millimeter wave radar devices and polysomnography.
Chest/abdominal movement and others | At baseline and millimeter wave radar monitoring or other devices continues during one month's or one year's follow-up
  Changes in chest/abdominal movement based on charts or indices and other non-specific measures will be monitored by millimeter wave radar devices or other devices.
Diagnosis of COPD according to lung function | At baseline
  The diagnosis of COPD is made according to the lung function criteria: post-bronchodilator FEV1 (forced expiratory volume at one second): FVC (forced vital capacity) less than 70%.
Diagnosis of sleep apnea hypopnea syndrome according to the times of apnea and hypopnea or AHI (RDI) with certain symptoms | At baseline
  The diagnosis of sleep apnea hypopnea syndrome is made according to the times of apnea and hypopnea more than 30 during 7-hour's sleep per night, or AHI is 5 times per hour or more (or using respiratory disturbance index if possible), with primarily obstructive apnea, snore, sleep apnea, and daytime sleepiness.

SECONDARY OUTCOMES:
The occurrence of acute exacerbation in patients with COPD combined with sleep apnea hypopnea syndrome | During one month's or one year's follow-up
  The occurrence of acute exacerbation in patients with COPD combined with sleep apnea hypopnea syndrome during follow-up
The time of occurrence of acute exacerbation in patients with COPD combined with sleep apnea hypopnea syndrome | During one month's or one year's follow-up
  The time of occurrence (from the prognosis data) of acute exacerbation in patients with COPD combined with sleep apnea hypopnea syndrome during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, Principal Investigator — Peking University Third Hospital
Locations (1):
- Tsinghua University, Beijing, China